CLINICAL TRIAL: NCT00032942
Title: A Phase III Placebo-Controlled, Double-Blind Multi-Site Trial of Lofexidine for Opiate Withdrawal
Brief Title: Lofexidine for Opiate Withdrawal - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Britannia Pharmaceuticals Ltd. (Industry)
Responsible Party: Ann Montgomery, National Institute on Drug about
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CSP-1020-1; NCT00007566 (obsolete NCT alias); NCT00024713 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-07

CONDITIONS: Opioid-Related Disorders
Keywords: opiate dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — lofexidine

INTERVENTIONS:
Drug: Lofexidine

SUMMARY:
The purpose of this study is to evaluate lofexidine for opiate withdrawal.

DETAILED DESCRIPTION:
An 11 day inpatient placebo-controlled, double-blind study of 96 opiate dependent, treatment seeking individuals randomized to 2 medication groups: lofexidine and placebo to be conducted in inpatient units at 3 treatment sites.

ELIGIBILITY:
Inclusion Criteria:

Male or female as least 18 yrs of age & above with a current dependence on heroin, morphine or hydromorphone according to DSM4 criteria; subject ; voluntarily given consent and signed informed consent; females using appropriate birth control method.

Exclusion Criteria:

Additional criteria available during screening at the site

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66
Dates: Start 2001-04; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Opiate withdrawal symptoms
Potential Abuse Liability

CONTACTS AND LOCATIONS:
Overall Officials: Ann Montgomery, R.N., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (3):
- United States (3):
  - UCLA Medical Center, Los Angeles, California
  - Columbia University, New York, New York
  - Philadelphia Veterans Medical Center, Philadelphia, Pennsylvania